CLINICAL TRIAL: NCT02976441
Title: Feasibility of Autologous Stem Cell Collection and Reinfusion in Newly Diagnosed High Grade Gliomas
Brief Title: Autologous Stem Cell Collection and Reinfusion in Newly Diagnosed High Grade Gliomas
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Physician decided not to go through with study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-x135
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Astrocytoma; Brainstem Glioma; Ependymoma; Mixed Glioma; Oligodendroglioma; Optic Nerve Glioma
MeSH Terms: conditions — Astrocytoma; Ependymoma; Glioma; Oligodendroglioma; Optic Nerve Glioma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal RT, Temozolomide, Stem Cell Collection/Reinfusion (Experimental): * Autologous stem cell collection will be performed 1-4 days prior to initiating radiation therapy and temozolomide
  * Focal radiation therapy: standard of care dose daily for approximately 6 weeks
  * Temozolomide: standard of care dose by mouth daily for 6 weeks with radiation
  * 2-7 days after the end of the radiation therapy and temozolomide the stem cells will be reinfused into the patient
  * Temozolomide: standard of care dose by mouth on days 1-5 every 28 days for 6 months following a 4-6 week rest period after the initial radiation and temozolomide
  Interventions: Radiation: Radiation therapy; Drug: Temozolomide; Procedure: Stem cell collection; Procedure: Stem cell infusion

INTERVENTIONS:
Radiation: Radiation therapy
Drug: Temozolomide
  Other Names: Temodar®
Procedure: Stem cell collection
Procedure: Stem cell infusion

SUMMARY:
The investigators hypothesize that this study will show that sufficient lymphocyte stem cell can be harvested prior chemoradiation and be reinfused back after treatment, and at least 5 of the 10 patients (50%) will achieve an absolute increase of lymphocyte counts of 300 cells/mm^3 four weeks after stem cell reinfusion in high grade glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed high grade glioma by pathology (WHO grade III or IV).
* At least 18 years of age.
* Karnofsky performance status ≥ 60%
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hematocrit ≥ 30%
  * Absolute lymphocyte count ≥ 1000/mcl Blood transfusions are permitted to allow potential participant to meet these criteria.
* Post-operative treatment plan must include standard radiation and temozolomide.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment with radiation therapy, chemotherapy, immunotherapy, biologic agents (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK, or gene therapy), or hormonal therapy. Glucocorticoid therapy is allowed.
* Anti-VEGF therapy within 6 weeks of registration.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any investigational agents that might affect lymphocytes. Patients receiving Novocure are allowed on study.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to filgrastim or plerixafor or other agents used in the study.
* Fresh CNS bleed as evident by MRI or CT.
* Contraindicated for anticoagulation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy of lymphocyte stem cell harvesting and reinfusion in patients as measured by the number of patients from whom 1-5x10e6 lymphocyte stem cells are collected and successfully reinfused without an adverse event | Completion of follow-up of all patients who received stem cell reinfusions (estimated to be 15 months)
  The study will provide preliminary evidence of efficacy if ≥5 of 10 patients (50%) achieve an increase over baseline in absolute lymphocyte counts (ALC) ≥300 cells/mm3 at 4 weeks after reinfusion from their baseline lymphocyte counts.

SECONDARY OUTCOMES:
Number of lymphocyte stem cells that can be harvested from this patient population | Completion of follow-up of all patients who received stem cell reinfusions (estimated to be 15 months)
Proportion of patients who have an increase in lymphocyte of ≥300 cells/mm^3 after autologous stem cell reinfusion. | 4 weeks after stem cell reinfusion
Duration of lymphocyte rise following stem cell reinfusion | Up to 6 months after stem cell reinfusion (approximately 9 months)
Changes in lymphocyte subtypes following collection and reinfusion | Up to 6 months after stem cell reinfusion (approximately 9 months)
  Lymphocyte subtypes will be monitored by flow cytometry at the time of stem cell collection, prior to autologous stem cell reinfusion, and then monthly for 6 months.
Changes in series of cytokine levels following collection and reinfusion | Up to 6 months after stem cell reinfusion (approximately 9 months)
  Cytokine levels will be checked by ELISPOT at the time of stem cell collection, weekly during radiation therapy/temozolomide (up to 6 weeks), prior to autologous stem cell reinfusion, and then monthly for 6 months.
Safety and toxicities with stem cell collection and reinfusion as measured by grade and frequency of adverse events | Up to 6 months after stem cell reinfusion (approximately 9 months)
  the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all adverse event/toxicity reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li Campian, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu